CLINICAL TRIAL: NCT00433134
Title: Survey Investigation of Adherence to Immunosuppression and Other Medications Among Kidney Transplant Recipients at SUNY Downstate
Brief Title: Survey of Adherence to Immunosuppression and Other Medications in Kidney Transplant Patients
Status: Completed | Type: Observational
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Mariana Markell, MD, SUNY Downstate MC
Other Study IDs: 06-093
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Last update posted 2009-04-24 (Estimated); Status verified 2009-04

CONDITIONS: Kidney Transplantation; Treatment Refusal; Patient Compliance
Keywords: renal transplant recipient; adherence; compliance; immunosuppression
MeSH Terms: conditions — Treatment Refusal; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Adherence

SUMMARY:
Goal:

To define the causes and issues associated with nonadherence in our population

Hypothesis:

There is a difference in the rates and patterns of adherence to transplant medications versus other medications also taken by transplant patients

Methods:

1. A standardized interviewer-administered confidential survey exploring levels of adherence to transplant medications and other medications as well questionnaires on a variety of cognitive and other factors known to be associated with adherence.
2. A brief review of demographics and pertinent laboratory information at the same encounter

DETAILED DESCRIPTION:
Objectives:

1. To determine the prevalence of nonadherence in our population
2. To assess possible causes of nonadherence and correlate those causes with demographic information and clinical findings
3. To assess for differences between adherence with immunosuppressive regime versus adherence with other medications (for hypertension, diabetes, hypercholesterolemia)

Methods:

1. A standardized interviewer-administered confidential survey exploring levels of adherence to transplant medications and other medications as well questionnaires on a variety of cognitive and other factors known to be associated with adherence
2. A brief review of demographics and pertinent laboratory information at the same encounter

ELIGIBILITY:
Inclusion Criteria:

* All renal transplant recipients with a working transplant who are currently attending the transplant clinic and who have been transplanted 6 months to 4.5 years ago are eligible. Patients are recruited at random from the transplant clinic waiting area

Exclusion Criteria:

* Less than 6 months post-transplant
* More than 4.5 years post transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Markell, MD, Principal Investigator — State University of New York - Downstate Medical Center; Sima Terebelo, MPH, RPA-C, Principal Investigator — State University of New York - Downstate Medical Center
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States